CLINICAL TRIAL: NCT00288093
Title: A Phase I Study of Triapine® in Combination With Radiation Therapy in Locally Advanced Pancreas Cancer
Brief Title: 3-AP and Radiation Therapy in Treating Patients With Stage III Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00120; NCI-2009-00120 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 05011; OSU-2005C0030; CSU-05011; CDR0000455065; NCI-7044; 05011 (Other: Ohio State University Comprehensive Cancer Center); 7044 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — Radiotherapy, Conformal; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Treatment (triapine, radiation therapy) (Experimental): Patients undergo radiotherapy once daily, 5 days a week, for approximately 5.5 weeks (a total of 28 fractions). Patients also receive 3-AP (Triapine) IV over 2 hours 3 days a week every other week for 5.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of 3-AP (Triapine) until the maximum tolerated dose (MTD) is determined.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Triapine

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy
Drug: Triapine

SUMMARY:
This phase I trial is studying the side effects and best dose of 3-AP when given together with radiation therapy in treating patients with stage III pancreatic cancer that cannot be removed by surgery.

3-AP may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. 3-AP may make tumor cells more sensitive to radiation therapy. Giving 3-AP together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerable dose (MTD) of 3-AP administered in combination with radiation therapy (XRT) in patients with locally advanced pancreatic carcinomas.

SECONDARY OBJECTIVES:

I. To document the therapeutic response of this combination in patients with locally advanced pancreatic carcinomas.

II. To establish radiographic correlates using secretin stimulated magnetic resonance cholangiopancreatography (MRCP) and dynamic contrast enhanced magnetic resonance imaging (MRI).

III. To measure deoxycytidine triphosphate (dCTP) levels in peripheral blood mononuclear cells (PBMCs)before and after treatment at specified times and try to correlate findings to activity and toxicity of triapine.

OUTLINE: This is a dose-escalation study of 3-AP (Triapine®). Patients undergo radiotherapy once daily, 5 days a week, for approximately 5½ weeks (a total of 28 fractions).

Patients also receive 3-AP (Triapine®) IV over 2 hours 3 days a week every other week for 5½ weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of 3-AP (Triapine®) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD. After completion of study treatment, patients are followed monthly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Unresectable nonmetastatic (stage III) disease
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST/ALT ≤ 3 times ULN
* Creatinine normal ORcreatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to 3-AP (Triapine®) or other agents used in study
* No known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would complicate compliance with study treatment
* No pulmonary disease (i.e., dyspnea at rest, requiring supplemental oxygen, or baseline oxygen saturation < 92%)
* No prior chemotherapy or radiotherapy
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12-20 (Actual); Primary Completion 2012-12-28 (Actual); Study Completion 2012-12-28 (Actual)

PRIMARY OUTCOMES:
MTD as assessed by the number of patients with dose-limiting toxicity (DLT) | Observed clinically for 3-4 hours after each 3-AP infusion during the first week of treatment
  MTD will be the dose at which 1 or fewer patients (less than or equal to 1/6) experiences a DLT during the treatment cycle with the next higher dose having at least 2/3 or 2/6 patients experiencing DLT. DLT will be defined as greater than or equal to Grade 3 non-hematologic or greater than or equal to Grade 4 hematologic adverse event with the following exceptions: greater than or equal to Grade 3 nausea and greater than or equal to Grade 3 vomiting that improves with antiemetic therapy greater than or equal to Grade 3 diarrhea that improves with Lomotil.

SECONDARY OUTCOMES:
Levels of dCTP in PBMCs correlated to activity and toxicity of 3-AP | Immediately before and after 3-AP on the first and last day of treatment
  The effect of 3-AP on dCTP levels in PBMCs will be evaluated using either a paired t-test or its nonparametric equivalent, the Wilcoxon matched pairs signed ranks test. Assuming normality, a paired t-test will allow us to detect an effect size of approximately 1.0 or greater in a sample of 12 patients with a two-sided alpha of 0.05 and a power of 0.88. All patients in a cohort will undergo the full 5 ½ weeks of therapy for toxicity assessment. NCI Common Toxicity Criteria version 4.0 will be used to grade toxicity.
Radiographic correlates using secretin-stimulated MRCP and dynamic contrast enhanced MRI | Prior to treatment (baseline), 2 weeks within and 4 weeks after combined-modality therapy
  The subjects will be imaged with conventional T2- and T1-weighted sequences prior to contrast agent application and with T1-weighted sequences after contrast agent application for tumor localization and volumetry. Dynamic contrast enhanced (DCE) images will be acquired to demonstrate tumor heterogeneity, microcirculation, vascularization and viability. Secretin-stimulated images will be acquired to quantify the functional status of the pancreas. The results will be purely descriptive.
Therapeutic response as assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) | CT scans at baseline and 4 weeks from end of therapy and then every 2 months for 1 year from start of therapy. Confirmatory scans will also be obtained 2 months following initial documentation of an objective response.
  Complete Response (CR) is the disappearance of all target lesions. Partial Response (PR) requires at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. The results will be purely descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States